CLINICAL TRIAL: NCT04500119
Title: Neuronal Mechanisms of Human Episodic Memory
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Johns Hopkins University (Other); University of Colorado, Denver (Other); University Health Network, Toronto (Other); Boston Children's Hospital (Other); University of California, Santa Barbara (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); California Institute of Technology (Other)
Responsible Party: Principal Investigator, Adam Mamelak, MD, Professor of Neurosurgery, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000572; 5U01NS117839-03 (NIH)
Record Dates: First submitted 2020-07-29; First posted 2020-08-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy Intractable
Keywords: Epilepsy; Decision-making; Memory; Depth Electrode
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Testing (Experimental): Behavioral and Neuronal Recordings
  Interventions: Behavioral: Cedrus RB-844 response pad; Adtech Behnke-Fried micro-electrodes; Neurolynx electrophysiology system; Blackrock Cerestim stimulator

INTERVENTIONS:
Behavioral: Cedrus RB-844 response pad; Adtech Behnke-Fried micro-electrodes; Neurolynx electrophysiology system; Blackrock Cerestim stimulator — Devices listed are components of a single intervention that includes: Record patient responses (Cedrus RB-844), record neuronal activity (Neurolynx) from electrodes (Adtech Behnke-Fried), apply intermittent electrical stimulation (Blackrock Cerestim)

SUMMARY:
The purpose the research is to better understand how the human brain accomplishes the basic cognitive tasks of learning new information, recalling stored information, and making decisions or choices about presented information. These investigations are critical to better understand human cognition and to design treatments for disorders of learning and memory.

DETAILED DESCRIPTION:
The rapid formation of new memories and the recall of old memories to inform decisions is essential for human cognition, but the underlying neural mechanisms remain poorly understood. The long-term goal of this research is a circuit-level understanding of human memory to enable the development of new treatments for the devastating effects of memory disorders. The study experiments utilize the rare opportunity to record in-vivo from human single neurons simultaneously in multiple brain areas in patients undergoing treatment for drug resistant epilepsy. The overall objective is to continue and expand a multi-institutional (Cedars Sinai/Caltech, Johns Hopkins, U Toronto, Children's/Harvard, UC Denver, UCSB), integrated, and multi-disciplinary team. Jointly, the investigators have the expertise and patient volume to test key predictions on the neural substrate of human memory. The study will utilize a combination of (i) in-vivo recordings in awake behaving humans assessing memory strength through confidence ratings, (ii) focal electrical stimulation to test causality, and (iii) computational analysis and modeling.

These techniques will be applied to investigate three overarching hypotheses on the mechanisms of episodic memory. First, to determine the role of persistent neuronal activity in translating working memories into longterm declarative memories (Aim 1). Second, to determine how declarative memories are translated into decisions (Aim 2). Third, to investigate how event segmentation, temporal binding and reinstatement during temporally extended experience facilitate episodic memory.

The expected outcomes of this work are an unprecedented characterization of how episodic memories are formed, retrieved and used for decisions, and how temporally extended experiences are segmented to form distinct but linked episodes. This work is significant because it moves beyond a "parts list" of neurons and brain areas by testing circuit-based hypotheses by simultaneously recording single-neurons from multiple frontal cortical and subcortical temporal lobe areas in humans who are forming, declaring and describing their memories. The proposed work is unusually innovative because it combines single-neuron recordings in multiple areas in behaving humans, develops new methods for non-invasive localization of implanted electrodes and electrical stimulation and directly test long-standing theoretical predictions on the role of evidence accumulation in memory retrieval.

A second significant innovation is the study team, which combines the patient volume and expertise of several major centers to maximally utilize the rare neurosurgical opportunities available to directly study the human nervous system. This innovative approach permits investigation of circuit-level mechanisms of human memory that cannot be studied non-invasively in humans nor in animal models. This integrated multi-disciplinary combination of human in-vivo single-neuron physiology, behavior, and modeling will contribute significantly to the understanding of the circuits and patterns of neural activity that give rise to human memory, which is a central goal of human neuroscience in general and the BRAIN initiative in particular.

ELIGIBILITY:
Inclusion Criteria:

* Intractable epilepsy, undergoing invasive monitoring
* Age ≥13
* Full Scale Intelligence Quotient > 70
* Ability to comprehend and perform simple behavioral tasks by pressing buttons on laptop computer in response to questions.

Exclusion Criteria:

* Determination by clinicians and investigators that a patient is unable to complete the behavioral tasks required for the protocol due to either cognitive limits, psychological limits, or pain.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Persistent Neuronal Activity (Firing Rates) | 3 years
  Neuronal firing rates (measured in spike rates per second) of cells in the frontal and temporal lobes during working memory.
Persistent Neuronal Activity (Power) | 3 years
  Power of local field potential bandwidths (measured in amplitude across frequency of the bandwidths) in the frontal and temporal lobes during working memory.
Decision Making (Firing Rates) | 5 years
  Neuronal firing rates of cells (measured in spike rates per second) in the frontal and temporal lobes during a decision-making process.
Decision Making (Power) | 5 years
  Power of local field potential bandwidths (measured in amplitude across frequency of the bandwidths) in the frontal and temporal lobes during a decision-making process.
Decision Making (Timing) | 5 years
  Timing of neuronal discharges (measured in spike rates per second) across the frontal and temporal lobes during a decision-making process.
Disruption of learning and memory via electrical stimulation (firing rates) | 5 years
  Measure the change in firing rates of neurons (measured in amplitude across frequency of the bandwidths) after applying small pulse of electrical activity during a learning task.
Disruption of learning and memory via electrical stimulation (memory) | 5 years
  Measure the change in memory (measured in spike rates per second) observed after applying small pulse of electrical activity during a learning task.

CONTACTS AND LOCATIONS:
Overall Officials: Ueli Rutishauser, PhD, Principal Investigator — Cedars-Sinai Medical Center; Adam Mamelak, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No